CLINICAL TRIAL: NCT01409655
Title: Centralized Off-Site Adherence Enhancement Program
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Yale University (Other); Harbor Medical Inc. (Industry)
Responsible Party: Principal Investigator, Honghu Liu, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R34DA031643 (NIH)
Record Dates: First submitted 2011-07-26; First posted 2011-08-04 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: HIV/AIDS, Medication Adherence
Keywords: AIDS, HIV, Adherence, Compliance, Contingency management
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Patient Compliance | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cognitive-behavioral therapy intervention (Experimental): Reinforcement for medication-taking will be wired to debit cards that patients will be given to receive the payments. This contingent reinforcement of medication-taking will be coupled with twelve sessions of cognitive-behavioral therapy (CBT) conducted by phone, also assisted by the website which will generate CBT-related text messages, reminders and scheduling information from a menu of choices negotiated by the patient and therapist.
  Interventions: Behavioral: cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: cognitive-behavioral therapy — . Reinforcement for medication-taking will be wired to debit cards that patients will be given to receive the payments. This contingent reinforcement of medication-taking will be coupled with twelve sessions of cognitive-behavioral therapy (CBT) conducted by phone, also assisted by the website which will generate CBT-related text messages, reminders and scheduling information from a menu of choices negotiated by the patient and therapist.
  Other Names: CARE

SUMMARY:
Our proposal "Centralized Off-Site Adherence Enhancement Program" or "CARE" will develop and test an effective behavioral adherence intervention program for HIV patients with alcohol and/or substance abuse problems. This project will develop and pilot test a novel program to help patients with alcohol and/or substance abuse problems take their medications as prescribed. The intervention will be delivered by phone, and utilize electronic monitoring of medication-taking, so patients can be treated by therapists from any geographic distance. To safely monitor data collected for this study, we have laid out a detailed Data Safety Monitoring Plan, which will cover all the issues required by NIDA.

DETAILED DESCRIPTION:
Patients who use drugs or alcohol who do not adequately adhere to antiretroviral medication have sub-optimal outcomes, but effective interventions for them are lacking. In this R34 application, we seek to develop and pilot an intervention program delivered by phone and supported by information technology that combines contingency management for medication adherence and a cognitive-behavioral approach to both adherence to antiretroviral therapy and abstinence from substances of abuse. The intervention, CARE (Centralized Off-site AdheRence Enhancement Program), builds on the published finding that adherence was robustly improved and viral load was significantly reduced among patients who received cash-reinforcement for opening MEMS-capped bottles to take prescribed medication on time. CARE involves transmission of bottle-opening data with real time operation from SimPill bottles to a website system which generates messages to patients indicating the amount of cash-reinforcement earned if medication was taken within a specified time window or forsaken if medication was missed. Reinforcement for medication-taking will be wired to debit cards that patients will be given to receive the payments. This contingent reinforcement of medication-taking will be coupled with twelve sessions of cognitive-behavioral therapy (CBT) conducted by phone, also assisted by the website which will generate CBT-related text messages, reminders and scheduling information from a menu of choices negotiated by the patient and therapist. Development of CARE will proceed in three stages, with revisions of the intervention at each stage. First, the web system and therapy manuals will be developed. Second, twelve weeks of CARE will be pre-piloted in 10 patients with sub-optimal adherence and recent risky alcohol use and/or stimulant misuse. Qualitative and quantitative data will be collected concerning acceptability, usability and perceived efficacy of components of CARE; Procedures and logistics will be evaluated, and modified, if necessary. Third, CARE will be pilot-tested in a twelve-week randomized controlled trial in which the control arm only involves phone-based counseling focusing first on adherence and then on abstinence. Retention of effects will be examined during a twelve-week follow-up period. CARE has the potential to be among the first interventions that delivers both reinforcement and counseling remotely, that improves outcomes among substance users without providing opioid substitution or other extremely intensive interventions, and that utilizes a cognitive-behavioral approach targeting both non-adherence and substance abuse. Because CARE is delivered by a therapist who is off-site from the patient's clinic, CARE can be effectively delivered from any distance and is a scalable treatment for patients in whom medication adherence is crucial.

ELIGIBILITY:
Inclusion Criteria:

* Current treatment with antiretroviral medications
* Within the last sixty days, either (a) Self-reported risky alcohol use (defined as >14 drinks/week or >4 drinks/occasion for men 65 or younger; >7 drinks/week or >3 drinks/occasion for women); OR (b) >=two days of either cocaine or amphetamine use
* Able to provide voluntary informed consent as evidenced by ability to answer questions about the consent form
* Able and willing to use SimPill caps to store at least one antiretroviral medication

Exclusion Criteria:

* Physiological dependence on alcohol, illicit opioids or sedatives as assessed by the history and symptom review procedures
* Dispensed medications in a monitored setting
* Unable to speak English. The need for bilingual staff and cross-coverage to enroll monolingual Hispanic people is beyond this study's scope.
* Will not be able to complete the study because of anticipated incarceration or move

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
change of adherence to antiretroviral medications measured at weeks 0, 4, 8, 12, 16, 20, and 24 | weeks 0, 4, 8, 12, 16, 20, and 24.
  collect information about adherence and behaviroal measures

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States